CLINICAL TRIAL: NCT04081441
Title: Impacts of Clean Cookstoves/Efficient Fuels Uptake and Empowerment Trainings on Women's Health and Well Being in Humanitarian Settings in Rwanda
Brief Title: Impacts of Clean Cookstoves and Empowerment Training on Women's Health in Refugee Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Fundacion Plan International Espana (Unknown); Global Alliance for Clean Cookstoves (Other); World Bank (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 7806
Record Dates: First submitted 2019-08-05; First posted 2019-09-09 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Gender-based Violence; Adherence; Mental Health Wellness 1; Empowerment; Food Insecurity; Relationship, Family
Keywords: gender-based violence; intimate-partner violence; empowerment; food insecurity; humanitarian settings; depression; fuel use; clean cookstoves
MeSH Terms: conditions — Empowerment; Depression

STUDY DESIGN:
Intervention Model Description: In this natural experiment, we have two connected randomized intervention deployments. The cookstove/fuel program was randomly rolled out to 750 households in Kigeme camp over a 6-month period (September 2018-March 2019) by Inyenyeri (a Rwandan social business). A second intervention (I-ACT empowerment training) was rolled out by Plan, International (December 2018-March 2019). I-ACT was deployed to women and their male partners (if applicable and available). After March 2019, the cookstove/pellet program was available to the whole camp. Assessments of impacts are done at 6 months after deployment of the interventions. Due to the staggering of the intervention roll-outs, the midline follow-up includes a six-month follow-up of the cookstove deployment and approximately 2-3 months of the I-ACT intervention and includes both partnered and non-partnered women. The 12-month assessment includes a 6-month follow up of the I-ACT empowerment intervention for partnered women only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Inyenyeri clean cookstove/fuel (Experimental): A tier 4 clean Mimi-moto cookstove/pellet system
  Interventions: Device: Inyenyeri clean cookstove and fuel system
- I-ACT behavioral empowerment intervention (Experimental): A culturally adapted 2-day personal empowerment workshop (based on the Individual, Agency-Centered Training (I-ACT) to women and modified, condensed 1-day training for their male partners, if applicable
  Interventions: Behavioral: I-ACT (Individual, Agency-Centered Training) workshop
- Cookstove and I-ACT empowerment (Experimental): Access to both the clean cookstove system and I-ACT empowerment training
  Interventions: Device: Inyenyeri clean cookstove and fuel system; Behavioral: I-ACT (Individual, Agency-Centered Training) workshop
- I-ACT Waitlisted control (Other): These households include those that were offered cookstoves after 6 months (from baseline) and are waitlisted to receive the I-ACT intervention
  Interventions: Device: Inyenyeri clean cookstove and fuel system

INTERVENTIONS:
Device: Inyenyeri clean cookstove and fuel system — The Inyenyeri cooking systems includes a tier 4 clean cooking system with biomass pellets that are purchased through the unconditional cash transfer program in the refugee camp
  Arms: Cookstove and I-ACT empowerment; I-ACT Waitlisted control; Inyenyeri clean cookstove/fuel
Behavioral: I-ACT (Individual, Agency-Centered Training) workshop — The I-ACT (Individual, Agency-Centered Training) empowerment workshop consists of behavioral exercises drawn primarily from positive psychology, that provide the tools to foster a growth mindset by allowing participants to understand the link between their thoughts, beliefs, and past actions to their future actions. Conducted in a workshop setting, this locally adapted version of the I-ACT curriculum consists of two days for women and a 1 day workshop for their male partners (as applicable)
  Arms: Cookstove and I-ACT empowerment; I-ACT behavioral empowerment intervention

SUMMARY:
The main objective of this study is to understand the links and outcomes of adoption of a cleaner cookstove/fuel and exposure to a personal empowerment training on women's health outcomes in a Congolese refugee camp in Rwanda, with a focus on gender-based violence (GBV).

DETAILED DESCRIPTION:
This randomized controlled trial examines the impacts of a phased-in integrated technology -behavior change intervention on women's health with a focus on gender-based violence. In a population of approximately 1500 Congolese households in Kigeme refugee camp in Rwanda, two interventions are randomly deployed in the camp. The first intervention is the Inyenyeri cookstove/pellet fuel system, a Tier 4 clean cookstove system; the second intervention is a behavior change intervention (referred to as I-ACT, Individual-Agency-Centered Training) designed to foster personal agency and empowerment, given to women and, if applicable, their male partner. Analyses will be done with interviews on 1500 women (ages 18-45) from these households that may have received one, both or none of the interventions, either as the full sample or the sub-sample of partnered-only women.

ELIGIBILITY:
Inclusion Criteria:

* Study participants are between the ages of 18 years - 45 years of age
* Reported as currently living in a refugee camp with no intention to relocate
* Has lived in any refugee camp for at least 1 year and can be interviewed in private
* Has the ability to give informed consent

Exclusion Criteria:

* Inability to provide informed consent
* Individuals having evidence of significant illness and/or are not able to engage fully in the surveys
* Women younger than 18 or over 45 years of age
* Those who have not lived continuously in a refugee camp setting for the past 12 months
* If two or more women live in a household, only one of these will be included in the study. The one responsible for fuel purchase/collection will be selected. If more than one woman is responsible for fuel collection, we will randomly choose one woman to participate in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 1555 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Rates of gender-based violence | 6 months
  Change in gender-based violence (GBV) over time as assessed through an adapted ASIST-GBV screening tool to identify physical violence, sexual violence, harassment, emotional violence and reproductive coercion between non-partners and intimate partners in humanitarian settings.
Number of households reporting uptake and consistent use of clean cooking system and fuel | 6 months
  Change in uptake and use of the clean cooking system as measured through pellet purchase and reported pellet use behavior
Number of participants reporting minor psychiatric disorders | 6 months
  Changes in the number of participants reporting minor psychiatric disorders as determined by the General Health Questionnaire (GHQ-12) as a result of the empowerment intervention.
Number of participants reporting anxiety and depression | 6 months
  Changes in the number of participants reporting anxiety and depression as determined by the Hopkins Symptom Checklist (HSCL) as a result of the empowerment intervention.
Number of participants reporting emotional symptoms of trauma | 6 months
  Changes in the number of participants reporting emotional symptoms of trauma as determined by the Harvard Trauma Questionnaire (HTQ) as a result of the empowerment intervention.
Number of participants reporting increased economic and social empowerment | 6 months
  Change in rates of reported uptake of economic activities (such as small businesses or savings) as well as participation in social groups and local training programs
Number of participants reporting reduced food insecurity | 6 months
  Change in reported incidence and severity of food insecurity as determined through a culturally adapted modification of the food insecurity experience scale (FIES) associated with food-related distress during the past month
Number of participants reporting increased self-efficacy | 6 months
  Changes in self-efficacy (as assessed by the New General Self-Efficacy Scale) as a result of the empowerment intervention.
Number of participants reporting increased grit | 6 months
  Changes in grit (Grit scale (Duckworth, et al)) as a result of the empowerment intervention.
Number of participants reporting increased social agency | 6 months
  Changes in social agency (as assessed by Ryff's psychological well-being scales) as a result of the empowerment intervention.

SECONDARY OUTCOMES:
Number of participants reporting increased quality and quantity of social networks | 6 months
  Changes in quality of social networks in the form of network size, network density and stove homophily resulting from either the empowerment training or the improved cookstove program as determined by reported social ties and characteristics of those social ties.

CONTACTS AND LOCATIONS:
Overall Officials: Anita V Shankar, Ph.D., Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Naira Kalra, Ph.D., Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Plan International, Rwanda, Kacyiru, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from this sample on social networks will be shared with colleagues at Boston College
Supporting Information: Analytic Code
Time Frame: August 2019-January 2020

REFERENCES:
- [Derived] Kalra N, Habumugisha L, Shankar A. Impacts of an abbreviated personal agency training with refugee women and their male partners on economic empowerment, gender-based violence, and mental health: a randomized controlled trial in Rwanda. BMC Public Health. 2024 May 14;24(1):1306. doi: 10.1186/s12889-024-18780-8. PMID 38745312